CLINICAL TRIAL: NCT00536380
Title: A Study of the Efficacy, Safety, and Quality of Life (QOL) in Patients With Chronic Idiopathic Urticaria Dosed With AERIUS Tablets (Desloratadine 5 mg, 10 mg, or 20 mg Once Daily)
Brief Title: Study for the Treatment of Chronic Idiopathic Urticaria With High Doses of AERIUS (Desloratadine) (Study P04849)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04849
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Results first posted 2010-05-03 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — desloratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5-mg Desloratadine (Experimental): 5-mg Desloratadine once daily
  Interventions: Drug: 5-mg Desloratadine
- 10-mg Desloratadine (Experimental): 10-mg Desloratadine once daily
  Interventions: Drug: 10-mg Desloratadine
- 20-mg Desloratadine (Experimental): 20-mg Desloratadine once daily
  Interventions: Drug: 20-mg Desloratadine

INTERVENTIONS:
Drug: 5-mg Desloratadine — 5-mg desloratadine tablets, once daily for four weeks.
  Other Names: SCH 34117, Clarinex, Aerius
  Arms: 5-mg Desloratadine
Drug: 10-mg Desloratadine — 10-mg desloratadine tablets, once daily for four weeks.
  Other Names: SCH 34117, Clarinex, Aerius
  Arms: 10-mg Desloratadine
Drug: 20-mg Desloratadine — 20-mg desloratadine tablets, once daily for four weeks.
  Other Names: SCH 34117, Clarinex, Aerius
  Arms: 20-mg Desloratadine

SUMMARY:
This study will investigate the effectiveness of desloratadine at doses higher (10 mg and 20 mg) than currently approved (5 mg) for the treatment of chronic idiopathic urticaria. Subjects with chronic urticaria who are currently taking a second generation antihistamine will be treated with desloratadine (5, 10, or 20 mg) for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria before being enrolled/randomized into the study.
* Subject must demonstrate willingness to participate in the study.
* Subject must be 18 to 75 years of age, of either gender, and any race.
* Subject must have had this episode of chronic idiopathic urticaria for at least 6 weeks or more, and has been dosing with a "2nd generation antihistamine (AH)" for 2 weeks or longer, and
* Subject's current episode of urticaria is sufficiently symptomatic at the Screening Visit to qualify for this study, in the opinion of the investigator.
* Subject has a Baseline Week (entry period) UAS between 10 and 30 inclusive.
* Patient must understand and be willing to assess and record symptom scores.
* Has voluntarily signed a written informed consent.
* Subjects must confirm that all prior medication washout times have been observed.
* Subject must confirm that he/she is practicing adequate contraception:

Female volunteers of childbearing potential (including women who are less than 1 year postmenopausal and women who will be sexually active during the study) must agree to use a medically accepted method of contraception or be surgically sterilized prior to screening, while receiving protocol-specified medication, and for 30 days after stopping the medication. Women who are postmenopausal for >1 year (i.e., women who have experienced 12 consecutive months of amenorrhea) will be exempted from the use of contraception during the study. Nonsterile or premenopausal female subjects must be using a medically accepted method of birth control, ie, double-barrier method (eg, male or female condom and spermicide), oral contraceptive, Depo-Provera, NuvaRing, contraceptive transdermal patch, etc, for female subjects of childbearing potential prior to screening and during the study. Women of childbearing potential should be counseled in the appropriate use of birth control while in the study. Vasectomy or tubal ligation is considered a single barrier. Women who are not currently sexually active must agree and consent to use one of the above-mentioned methods if they become sexually active while participating in the study.

* If subject is a female volunteer of childbearing potential, she must have a negative urine pregnancy test at Screening/Visit 1.
* Subjects must be free of any clinically relevant disease other than chronic idiopathic urticaria (CIU) that would, in the principal investigator's and/or sponsor's opinion, interfere with the conduct of the study or study evaluations.
* Subjects must be able to adhere to the dosing and visit schedules and agree to record symptom severity scores, medication times, concomitant medications, and adverse events (AEs) accurately and consistently in a daily diary.

Exclusion Criteria:

* Is a female who is pregnant, or intends to become pregnant during the study.
* Is nursing, or intends to be nursing during the study or within 90 days after study completion.
* Has not observed the designated washout periods for any of the prohibited medications.
* Has used any investigational product within 30 days prior to enrollment.
* Have any of the following clinical conditions:

  * Symptomatic seasonal or perennial allergic rhinitis.
  * Asthma not controlled by short-acting beta-2 agonists used as necessary.
  * The presence of permanent severe diseases, especially those affecting the immune system, except urticaria.
  * The presence of a permanent gastrointestinal condition which may influence the oral therapy (chronic diarrhea diseases, congenital malformations or surgical mutilations of gastrointestinal tract).
  * History of/or presence of epilepsy, significant neurological disorders, cerebrovascular attacks or ischemia.
  * History of/or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy.
  * Evidence of/or a history of significant renal disease.
  * Evidence of/or a history of significant hepatic disease.
  * Presence of cancer which requires chemotherapy or radiation therapy.
  * Presence of glaucoma.
  * Presence of urinary bladder neck obstruction with emptying difficulties.
  * Presence of acute urticaria .
  * Body mass index (BMI) > 35
* Has any clinically significant deviation from the appropriate reference range in the physical examination, or other clinical evaluation that, in the investigator's judgment, may interfere with the study evaluation or affect subject safety.
* Is in a situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.
* Is participating in any other clinical study(ies).
* Is on the staff, affiliated with, or a family member of the staff personnel directly involved with this study.
* Is allergic to or has a history of hypersensitivity to the study drug (desloratadine), to any of its excipients, or to loratadine.
* Has the rare hereditary problem of galactose intolerance, the Lapp lactase deficiency, or glucose-galactose malabsorption.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2007-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 5-mg Desloratadine | 10-mg Desloratadine | 20-mg Desloratadine
Started | 106 | 104 | 104
Completed | 94 | 95 | 94
Not Completed | 12 | 9 | 10
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal unrelated to study drug | 2 | 0 | 1
Not completed — Withdrawal related to study drug | 7 | 5 | 2
Not completed — Noncompliance with protocol | 3 | 2 | 2
Not completed — Did not meet protocol eligibility | 0 | 0 | 1
Not completed — Administrative | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5-mg Desloratadine | 10-mg Desloratadine | 20-mg Desloratadine | Total
Number analyzed (Participants) | 106 | 104 | 104 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (12.8) | 40.4 (13.3) | 40.1 (14.2) | 40.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 70 | 209
  Male | 36 | 35 | 34 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in the Urticaria Activity Score (UAS) From Baseline to the Final Week for Desloratadine 5 mg Versus Desloratadine 20 mg
Description: The UAS is a composite diary-recorded score. The diary recorded scores included wheal score and pruritus score with numeric severity intensity ratings of 0 = none to 3 = intense. The scoring was to be done twice daily within one hour of arising and in the evening, approximately 12 hours later. Scoring was "reflective", covering the 12-hour period since the previous recording. The daily UAS is the average of the morning and evening scores. The final week by definition was the terminal week. It was the last week participants stayed for the treatment period.
Time Frame: Baseline and 4 treatment weeks
Population: Intent to treat population
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | 5-mg Desloratadine | 20-mg Desloratadine | 10-mg Desloratadine
Number analyzed (Participants) | 104 | 100 | 104
Units on a scale
  Change from Baseline in UAS | -1.0 (0.12) | -1.0 (0.12) | -1.1 (0.12)
  Baseline UAS (mean +/- standard deviation) | 2.9 (0.82) | 2.8 (0.74) | 2.9 (0.77)
Statistical Analysis 1: Comparison: 5-mg Desloratadine vs 20-mg Desloratadine; Test type: Superiority or Other; p = 0.721, ANCOVA

ADVERSE EVENTS:
Arm/Group | 5-mg Desloratadine | 10-mg Desloratadine | 20-mg Desloratadine
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/104 | 1/104
Other Adverse Events (participants affected / at risk) | 5/106 | 4/104 | 6/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Desloratadine (N=106) | 10-mg Desloratadine (N=104) | 20-mg Desloratadine (N=104)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-mg Desloratadine (N=106) | 10-mg Desloratadine (N=104) | 20-mg Desloratadine (N=104)
Headache (Nervous system disorders) | 5 (6) | 4 (5) | 6 (9)

LIMITATIONS AND CAVEATS:
Due to poor enrollment (even after extending the enrollment period), only 314 participants (not 600 participants) were randomized to the study and hence the study was inconclusive due to the lacking of statistical power and robustness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to publish or publicly present any interim results of Study without prior written consent of sponsor. PI further agrees to provide 45 days written notice to sponsor prior to submission for publication or presentation to permit sponsor to review copies of abstracts or manuscripts for publication (including, without limitation, slides and text of oral or other public presentations and text of any transmission through any electronic media) which report any results of Study.